CLINICAL TRIAL: NCT02179710
Title: Cystic Fibrosis Treatment Adherence Cayston Proof-of-Concept Pilot Study
Status: Completed | Type: Observational
Sponsor: Landon Pediatric Foundation (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: M.O.M.M.I.1; M.O.M.M.I.1 (Registry Identifier: M.O.M.M.I.PBRN)
Record Dates: First submitted 2014-06-30; First posted 2014-07-02 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Cystic Fibrosis
Keywords: adherence; cystic fibrosis; adolescents; adults
MeSH Terms: conditions — Cystic Fibrosis | interventions — Aztreonam

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Motivational Interviewing: Review of adherence dashboard by the investigator with the patient to facilitate and engage intrinsic motivation within the client in order to change behavior.
  Interventions: Behavioral: Adherence dashboard motivational interviewing

INTERVENTIONS:
Behavioral: Adherence dashboard motivational interviewing — These data will be aggregated and displayed graphically in weekly intervals. Adherence will be displayed as percentage and timing percentage within a set criterion of prescribed inter-dose interval. Drug holidays, operationally defined as missing two or more consecutive doses will be displayed along with average length. Patient self-reported adherence information, collected via handheld (i.e, smart phone, tablet, laptop) application will be displayed as percentage and timing percentage on the dashboard. Review of dashboard weekly with investigator for motivational interviewing
  Other Names: PARI; Altera; Cayston

SUMMARY:
Real-world adherence to inhaled and oral therapies for cystic fibrosis (CF) patients remains discouragingly low, ranging between 31-53% for inhaled antibiotics and 41-72% for hypertonic saline. Programs to enhance adherence, including comprehensive behavioral interventions with adolescents, have met with mixed success. Advances in therapy, treatment delivery systems, and data capture technology offer the potential for enhancing adherence by providing immediate and more frequent feedback to the patient regarding his or her fidelity to the prescribed treatment regimen. We propose to conduct a proof-of-concept study to evaluate a systematic approach to linking treatment and feedback components to enhance adherence.

DETAILED DESCRIPTION:
Study Design: This will be a single group intervention involving a 28-day baseline (Phase 1), a 28-day treatment period with enhanced adherence feedback. Subjects will be treated with Cayston via a blue tooth enabled nebulizer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be 18 non-adherent CF patients
* Stratified by age as adult supervised (8-12) adolescents (12-18) and young adults (19-30) and gender
* Balanced for ethnicity and disease severity -Non-adherence status will be determined at screening based on an MAQ score < 6. -

Exclusion Criteria:

* Inability to give informed consent or assent

Ages: 8 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with cystic fibrosis over age 8 with difficulties with adherence to aerosolized Caysotn
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2015-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Remotely Observed Therapy | 140 days
  Doses of medication as recorded by bluetooth device

SECONDARY OUTCOMES:
Morisky Adherence Questionnaire | 140 days
  Changes in self reported adherence

CONTACTS AND LOCATIONS:
Overall Officials: Chris Landon, MD, Principal Investigator — Landon Pediatric Foundation
Locations (1):
- Pediatric Diagnostic Center, Ventura, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Will be made available to other users of PARI blue tooth monitoring